CLINICAL TRIAL: NCT03098212
Title: Efficacy of Aromatherapy for Reducing Pain During Labor
Brief Title: Aromatherapy for Reducing Labor Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kuntharee Traisrisilp, Principle investigator, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3487
Record Dates: First submitted 2017-03-08; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Aromatherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy (Experimental): Receive essential oil diffuse by Aroma diffuser during labor. Pain score and dose of analgesics drug are recorded
  Interventions: Other: Aromatherapy
- Non-aromatherapy (No Intervention): This group receive pain control by standard of care without essential oil (aromatherapy)

INTERVENTIONS:
Other: Aromatherapy — On the day of admission for labor. Pregnant women select type of essential oil. Aroma diffuser is used during labor. Pain score was record during latent, early active and late active phase.
  Arms: Aromatherapy

SUMMARY:
Pregnant women who eligible with inclusion criteria are random to two groups. Aromatherapy group will receive the aromatherapy during labor along with standard pain control.

Non-aromatherapy group will receive standard pain control during labor

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Nulliparous
* 37 complete weeks of gestation
* Cephalic presentation
* No emergency obstetric complication
* In labor

Exclusion Criteria:

* Medical or obstetric complication preclude vaginal delivery
* Essential oil allergy
* Side effect of aromatherapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
early active phase pain using Visual Analog Scale | The day of labor
  Visual analog scale used to assess pain during cervical dilate 5-7 cm.

SECONDARY OUTCOMES:
latent phase pain using Visual Analog Scale | The day of labor
  Visual analog scale used to assess pain during cervical dilate 3-4 cm.
late active phase pain using Visual Analog Scale | The day of labor
  Visual analog scale used to assess pain during cervical dilate 8-10 cm.
analgesic drug | The day of labor
  doses of analgesic drug request by pregnant women

IPD SHARING:
Plan to Share IPD: No